CLINICAL TRIAL: NCT02084576
Title: Comparison of Ketorolac Tromethamine 0.4% and Nepafenac 0.1% for the Prevention of Cystoid Macular Edema After Phacoemulsification: Prospective Randomized Double-masked Study
Brief Title: Anti-inflammatory Efficacy for Prophylaxis of Cystoid Macular Edema (CME) After Phacoemulsification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Oftalmologico de Brasilia (Other)
Responsible Party: Principal Investigator, PATRICK FRENSEL DE MORAES TZELIKIS, Principal Investigator, Hospital Oftalmologico de Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014.02; HOB03022014 (Other: HOB-14/02)
Record Dates: First submitted 2014-02-18; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Cystoid Macular Edema; Cataract
Keywords: Cystoid macular edema; nonsteroidal anti-inflammatory drug; OCT; phacoemulsification.
MeSH Terms: conditions — Macular Edema; Cataract | interventions — nepafenac; Ketorolac

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nepafenac (Experimental): One drop in the study eye 3 times daily for 30 days
  Interventions: Drug: Nepafenac
- Ketorolac (Active Comparator): One drop in the study eye 4 times daily for 30 days
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Nepafenac — One drop in the study eye 3 times daily for 30 days
  Other Names: Nevanac
  Arms: Nepafenac
Drug: Ketorolac — One drop in the study eye 4 times daily for 30 days
  Other Names: Acular LS
  Arms: Ketorolac

SUMMARY:
To compare the anti-inflammatory efficacy of ketorolac of tromethamine 0.4% and nepafenac 0.1% eye drops for prophylaxis of cystoid macular edema (CME) after small-incision cataract extraction.

DETAILED DESCRIPTION:
This prospective randomized clinical trial study included patients older than 40 years with age-related cataract, and a normal ophthalmologic examination besides senile cataract. Exclusion criteria were previous ocular surgery, central endothelial cell count less than 2000 cells/mm2, glaucoma or intraocular pressure greater than 21 mmHg, amblyopia, retinal abnormalities, steroid or immunosuppressive treatment, connective tissue diseases, or an allergy or hypersensitivity to NSAIDs. Enrolled patients who had complicated cataract surgery (eg, posterior capsule rupture, vitreous loss, or an intraocular lens not placed in the capsular bag) were subsequently excluded.

Study Protocol Preoperatively, patients had an extensive ophthalmologic examination, including measurement of corrected distance visual acuity (CDVA), refraction, slitlamp examination, intraocular pressure (IOP), fundoscopy, corneal endothelial cell count by noncontact specular microscopy (Noncon Robo, Konan), central corneal thickness (CCT) measurement (Pentacam, Oculus, Inc.), and biometry with the IOLMaster partial coherence interferometry device (Carl Zeiss Meditec AG). The targeted postoperative refractive error was 0.0 D. The visual acuity measurements were recorded with logMAR UDVA and CDVA.

In addition, a baseline spectral-domain OCT (SD-OCT) scan was performed before surgery and postoperatively after 1, 4 and 12 weeks. All SD-OCT imaging was performed with a spectral-domain Heidelberg Spectralis OCT devise (Heidelberg Engineering, Inc., Heidelberg, Germany).

Patients were assigned in a 1:1 ration to 1 of 2 treatments groups using a computer-generated randomization list. The study medications were ketorolac tromethamine 0.4% (Acular LS, Allergan) in group 1, and nepafenac 0.1% (Nevanac, Alcon) in group 2. Patients were instructed to instill ketorolac tromethamine 0.4% 1 drop in the operative eye 4 times a day (breakfast, lunch, dinner, and before bedtime), and nepafenac 0.1% 1 drop 3 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years with age-related cataract, and a normal ophthalmologic examination besides senile cataract.

Exclusion Criteria:

* Previous ocular surgery, central endothelial cell count less than 2000 cells/mm2, glaucoma or intraocular pressure greater than 21 mmHg, amblyopia, retinal abnormalities, steroid or immunosuppressive treatment, connective tissue diseases, or an allergy or hypersensitivity to NSAIDs. Enrolled patients who had complicated cataract surgery (eg, posterior capsule rupture, vitreous loss, or an intraocular lens not placed in the capsular bag) were subsequently excluded

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The incidence of CME was evaluated by retinal foveal thickness on optical coherence tomography (OCT) | After 1 week, 4 weeks, 12 weeks after surgery

SECONDARY OUTCOMES:
Postoperative corrected distance visual acuity | 4 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F Tzelikis, MD, PhD, Principal Investigator — Hospital Oftalmologico de Brasilia
Locations (1):
- Hospital Oftalmologico de Brasília, Brasília, Federal District, Brazil

REFERENCES:
- [Result] Shelsta HN, Jampol LM. Pharmacologic therapy of pseudophakic cystoid macular edema: 2010 update. Retina. 2011 Jan;31(1):4-12. doi: 10.1097/IAE.0b013e3181fd9740. PMID 21187730
- [Result] Brar M, Yuson R, Kozak I, Mojana F, Cheng L, Bartsch DU, Oster SF, Freeman WR. Correlation between morphologic features on spectral-domain optical coherence tomography and angiographic leakage patterns in macular edema. Retina. 2010 Mar;30(3):383-9. doi: 10.1097/IAE.0b013e3181cd4803. PMID 20216291
- [Result] Almeida DR, Johnson D, Hollands H, Smallman D, Baxter S, Eng KT, Kratky V, ten Hove MW, Sharma S, El-Defrawy S. Effect of prophylactic nonsteroidal antiinflammatory drugs on cystoid macular edema assessed using optical coherence tomography quantification of total macular volume after cataract surgery. J Cataract Refract Surg. 2008 Jan;34(1):64-9. doi: 10.1016/j.jcrs.2007.08.034. PMID 18165083
- [Derived] Tzelikis PF, Vieira M, Hida WT, Motta AF, Nakano CT, Nakano EM, Alves MR. Comparison of ketorolac 0.4% and nepafenac 0.1% for the prevention of cystoid macular oedema after phacoemulsification: prospective placebo-controlled randomised study. Br J Ophthalmol. 2015 May;99(5):654-8. doi: 10.1136/bjophthalmol-2014-305803. Epub 2014 Nov 10. PMID 25385061